CLINICAL TRIAL: NCT03379025
Title: Effects of Electronic Cigarettes on Smokers With Mild to Moderate Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Electronic Cigarettes in Cigarette Smokers With Mild to Moderate COPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: did not start RCT due to current concerns about vaping-related lung illness
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sara Kalkhoran, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017P002418
Record Dates: First submitted 2017-12-08; First posted 2017-12-20 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: COPD; Tobacco Use
Keywords: electronic cigarettes; e-cigarettes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Tobacco Use; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intervention Group (Experimental): JUUL Electronic Cigarettes, nicotine concentration 59 mg/ml, to replace all cigarette use for 12 weeks
  Interventions: Other: Electronic cigarette
- Delayed Intervention Group (Other): After a 12 week period of no electronic cigarette use, JUUL Electronic Cigarettes, nicotine concentration 59 mg/ml, to replace all cigarette use for 12 weeks
  Interventions: Other: Electronic cigarette

INTERVENTIONS:
Other: Electronic cigarette — electronic cigarette and cartridge refills (also known as pods)
  Other Names: e-cigarette, JUUL electronic cigarette

SUMMARY:
This study evaluates the effects of electronic cigarette use on cigarette smoking and markers of tobacco use, as well as respiratory symptoms and function in smokers with mild to moderate chronic obstructive pulmonary disease (COPD). All participants will receive a 12 week supply of electronic cigarettes to use instead of their regular conventional cigarettes.

DETAILED DESCRIPTION:
Electronic cigarettes are devices that heat a solution containing nicotine to form an aerosol that is then inhaled by the user. Electronic cigarettes are used by many smokers, including smokers with chronic health conditions such as COPD. Given that e-cigarettes are still relatively new, their effects on health are not well defined.

It is important to understand how electronic cigarettes affects symptoms and lung function in smokers with COPD to determine the short-term safety of these products. To do this, an initial step involves observing the extent to which smokers substitute their conventional cigarette use with electronic cigarette use and change their exposure to tobacco use biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* At least 10 pack year smoking history
* Daily use of at least 5 cigarettes
* No plan to quit cigarettes in the next 30 days
* Willing to use e-cigarettes
* Diagnosis of COPD (FEV1/forced vital capacity [FVC] <0.70) with mild (FEV1 >80% predicted) or moderate (FEV1 <80% but >50% predicted) airflow limitation (post-bronchodilator); confirmed by spirometry
* English-speaking

Exclusion Criteria:

* Past 30-day use of nicotine-containing products (cigars, cigarillos, hookah, electronic cigarettes, smokeless tobacco, nicotine replacement therapy)
* Past 30 day use of inhaled drugs (marijuana, crack)
* Pregnant or breastfeeding
* Planning to become pregnant within the next 3 months or unable to agree to use appropriate contraception during study
* Pulmonary disease other than COPD or asthma
* Ever requiring mechanical ventilation
* 2 or more hospitalizations for COPD in the past 12 months
* Cardiac hospitalization in the past 6 months
* Active chest pain or palpitations
* Uncontrolled hypertension (blood pressure >160/100)
* Oxygen therapy
* Inability or contraindication to perform spirometry (e.g. recent eye, thoracic, or abdominal surgery)
* Known allergy to propylene glycol or vegetable glycerin
* Unable to consent or complete assessments

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in cigarettes per day | baseline and 12 weeks
  Change in self-reported cigarettes per day from Week 0 to Week 12

SECONDARY OUTCOMES:
Change in urine anabasine | baseline and 12 weeks
  Change in tobacco biomarker anabasine from Week 0 to Week 12
Change in urine cotinine | baseline and 12 weeks
  Change in nicotine metabolite cotinine from Week 0 to Week 12
Change in exhaled carbon monoxide | baseline and 12 weeks
  Change in exhaled carbon monoxide from Week 0 to Week 12
Change in pulmonary function | baseline and 12 weeks
  Change in post-bronchodilator forced expiratory volume in one second (FEV1) from Week 0 to Week 12
Transition Dyspnea Index | baseline and 12 weeks
  Change in Transition Dyspnea Index at Week 12 from the Baseline Dyspnea Index at Week 0
St. George's Respiratory Questionnaire | baseline and 12 weeks
  Change in quality of life as measured by the St. George's Respiratory Questionnaire from Week 0 to Week 12

OTHER OUTCOMES:
Sustained change in cigarettes per day | 12 weeks and 24 weeks for immediate intervention group; 24 weeks and 36 weeks for delayed intervention group
  Assess whether any changes in cigarettes per day after 12 weeks of receiving e-cigarettes are sustained after an additional 12 weeks
Sustained change in urine anabasine | 12 weeks and 24 weeks for immediate intervention group; 24 weeks and 36 weeks for delayed intervention group
  Assess whether any changes in urine anabasine after 12 weeks of receiving e-cigarettes are sustained after an additional 12 weeks
Sustained change in urine cotinine | 12 weeks and 24 weeks for immediate intervention group; 24 weeks and 36 weeks for delayed intervention group
  Assess whether any changes in urine cotinine after 12 weeks of receiving e-cigarettes are sustained after an additional 12 weeks
Sustained change in exhaled carbon monoxide | 12 weeks and 24 weeks for immediate intervention group; 24 weeks and 36 weeks for delayed intervention group
  Assess whether any changes in exhaled carbon monoxide after 12 weeks of receiving e-cigarettes are sustained after an additional 12 weeks
Sustained change in pulmonary function | 12 weeks and 24 weeks for immediate intervention group; 24 weeks and 36 weeks for delayed intervention group
  Assess whether any changes in post-bronchodilator FEV1 after 12 weeks of receiving e-cigarettes are sustained after an additional 12 weeks
Sustained change in transition dyspnea index | 12 weeks and 24 weeks for immediate intervention group; 24 weeks and 36 weeks for delayed intervention group
  Assess whether any changes in post-bronchodilator FEV1 after 12 weeks of receiving e-cigarettes are sustained after an additional 12 weeks
Sustained change in St. George's Respiratory Questionnaire | 12 weeks and 24 weeks for immediate intervention group; 24 weeks and 36 weeks for delayed intervention group
  Assess whether any changes in quality of life as measured by the St. George's Respiratory Questionnaire after 12 weeks of receiving e-cigarettes are sustained after an additional 12 weeks